CLINICAL TRIAL: NCT07206550
Title: The Role of Framing and Choice Architecture in Patients' Reactions and Electronic Health Records' Error Discovery and Reporting
Brief Title: The Role of Framing and Choice Architecture in Patients' Reactions and EHR Error Discovery and Reporting
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Dr. Ryan Raimi, Assistant Professor of Information Systems, The University of Texas at Dallas
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: IRB-26-19
Record Dates: First submitted 2025-09-18; First posted 2025-10-03 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Electronic Health Records
Keywords: Electronic Health Records; EHR error; error discovery; error reporting; patient portal

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Control group (No Intervention): The participants in this arm will not receive any message, encouraging them to review their EHRs and report any potential errors.
- Gain Framing x Egocentric x "Errors" (Active Comparator): The participants in this arm will receive the following message using the term "errors", encouraging them to review their EHRs and report any potential errors: "If you review your medical record, there is a 20% risk of having an error in your EHR. This is a great opportunity to act as your own best advocate, check your EHRs to identify any potential errors, and improve your health outcomes."
  Interventions: Behavioral: Framing
- Loss Framing x Egocentric x "Errors" (Active Comparator): The participants in this arm will receive the following message using the term "errors", encouraging them to review their EHRs and report any potential errors: "If you review your medical record, there is a 20% risk of having an error in your EHR. Taking no action could lead to severe health-related consequences and occasionally be deadly. Act now and save yourself from experiencing the preventable negative consequences of having a potential error in your EHR."
  Interventions: Behavioral: Framing
- Gain Framing x Allocentric x "Errors" (Active Comparator): The participants in this arm will receive the following message using the term "errors", encouraging them to review their EHRs and report any potential errors: "If you review your medical record, there is a 20% risk of having an error in your EHR. Such errors can also affect those close to us not just ourselves. This is a great opportunity to act in the interest of your loved ones by improving your health outcomes via checking your EHRs to identify any potential errors. Your loved ones will thank you for prioritizing your safety."
  Interventions: Behavioral: Framing
- Loss Framing x Allocentric x "Errors" (Active Comparator): The participants in this arm will receive the following message using the term "errors", encouraging them to review their EHRs and report any potential errors: "If you review your medical record, there is a 20% risk of having an error in your EHR. Such errors can also affect those close to us not just ourselves. Taking no action could lead to severe health-related consequences and occasionally be deadly. Act now and save your loved ones from experiencing the preventable negative consequences of having a potential error in your EHR. Your loved ones will thank you for prioritizing your safety."
  Interventions: Behavioral: Framing
- Gain Framing x Egocentric x "Unintended Mistakes" (Active Comparator): The participants in this arm will receive the following message using the term "unintended mistakes", encouraging them to review their EHRs and report any potential errors: "If you review your medical record, there is a 20% risk of having an unintended mistake in your EHR. This is a great opportunity to act as your own best advocate, check your EHRs to identify any potential unintended mistakes, and improve your health outcomes."
  Interventions: Behavioral: Framing
- Loss Framing x Egocentric x "Unintended Mistakes" (Active Comparator): The participants in this arm will receive the following message using the term "unintended mistakes", encouraging them to review their EHRs and report any potential errors: "If you review your medical record, there is a 20% risk of having an unintended mistake in your EHR. Taking no action could lead to severe health-related consequences and occasionally be deadly. Act now and save yourself from experiencing the preventable negative consequences of having a potential unintended mistake in your EHR."
  Interventions: Behavioral: Framing
- Gain Framing x Allocentric x "Unintended Mistakes" (Active Comparator): The participants in this arm will receive the following message using the term "unintended mistakes", encouraging them to review their EHRs and report any potential errors: "If you review your medical record, there is a 20% risk of having an unintended mistake in your EHR. Such unintended mistakes can also affect those close to us not just ourselves. This is a great opportunity to act in the interest of your loved ones by improving your health outcomes via checking your EHRs to identify any potential unintended mistakes. Your loved ones will thank you for prioritizing your safety."
  Interventions: Behavioral: Framing
- Loss Framing x Allocentric x "Unintended Mistakes" (Active Comparator): The participants in this arm will receive the following message using the term "unintended mistakes", encouraging them to review their EHRs and report any potential errors: "If you review your medical record, there is a 20% risk of having an unintended mistake in your EHR. Such unintended mistakes can also affect those close to us not just ourselves. Taking no action could lead to severe health-related consequences and occasionally be deadly. Act now and save your loved ones from experiencing the preventable negative consequences of having a potential unintended mistake in your EHR. Your loved ones will thank you for prioritizing your safety."
  Interventions: Behavioral: Framing
- Gain Framing x Egocentric x "Inaccuracies" (Active Comparator): The participants in this arm will receive the following message using the term "inaccuracies", encouraging them to review their EHRs and report any potential errors: "If you review your medical record, there is a 20% risk of having an inaccuracy in your EHR. This is a great opportunity to act as your own best advocate, check your EHRs to identify any potential inaccuracies, and improve your health outcomes."
  Interventions: Behavioral: Framing
- Loss Framing x Egocentric x "Inaccuracies" (Active Comparator): The participants in this arm will receive the following message using the term "inaccuracies", encouraging them to review their EHRs and report any potential errors: "If you review your medical record, there is a 20% risk of having an e inaccuracy in your EHR. Taking no action could lead to severe health-related consequences and occasionally be deadly. Act now and save yourself from experiencing the preventable negative consequences of having a potential inaccuracy in your EHR."
  Interventions: Behavioral: Framing
- Gain Framing x Allocentric x "Inaccuracies" (Active Comparator): The participants in this arm will receive the following message using the term "inaccuracies", encouraging them to review their EHRs and report any potential errors: "If you review your medical record, there is a 20% risk of having an inaccuracy in your EHR. Such inaccuracies can also affect those close to us not just ourselves. This is a great opportunity to act in the interest of your loved ones by improving your health outcomes via checking your EHRs to identify any potential inaccuracies. Your loved ones will thank you for prioritizing your safety."
  Interventions: Behavioral: Framing
- Loss Framing x Allocentric x "Inaccuracies" (Active Comparator): The participants in this arm will receive the following message using the term "inaccuracies", encouraging them to review their EHRs and report any potential errors: "If you review your medical record, there is a 20% risk of having an inaccuracy in your EHR. Such inaccuracies can also affect those close to us not just ourselves. Taking no action could lead to severe health-related consequences and occasionally be deadly. Act now and save your loved ones from experiencing the preventable negative consequences of having a potential inaccuracy in your EHR. Your loved ones will thank you for prioritizing your safety."
  Interventions: Behavioral: Framing

INTERVENTIONS:
Behavioral: Framing — The participants will receive different messages using different terms and behavioral framings, encouraging them to review their EHRs and report any potential errors. These wording variations are expected to induce variance in subjects' behaviors with regard to the likelihood of reviewing EHRs, as well as discovering and reporting potential errors in them.
  Arms: Gain Framing x Allocentric x "Errors"; Gain Framing x Allocentric x "Inaccuracies"; Gain Framing x Allocentric x "Unintended Mistakes"; Gain Framing x Egocentric x "Errors"; Gain Framing x Egocentric x "Inaccuracies"; Gain Framing x Egocentric x "Unintended Mistakes"; Loss Framing x Allocentric x "Errors"; Loss Framing x Allocentric x "Inaccuracies"; Loss Framing x Allocentric x "Unintended Mistakes"; Loss Framing x Egocentric x "Errors"; Loss Framing x Egocentric x "Inaccuracies"; Loss Framing x Egocentric x "Unintended Mistakes"

SUMMARY:
The first goal of our research is to understand the effects of different wordings of certain messages on patients' engagement in reviewing their electronic health records (EHRs). These messages will be about EHR errors and their potential consequences, as well as the benefits that might accrue from reviewing EHRs. The second goal is to understand the effects of different wordings of certain messages on patients' discovery and reporting of potential errors in their electronic health records (EHRs).

The main questions it aims to answer are:

1. Does focusing on the negative OR positive consequences of EHR errors in the investigator's messages to people, increase their likelihood of reviewing their EHRs?
2. Does focusing on the negative OR positive consequences of EHR errors in the investigators' messages to people, increase their likelihood of discovery and reporting of potential errors in their EHRs?

First, participants will take an initial short online survey (for about 5 minutes).

Next, participants will be asked to log into their patient portal and review their EHRs, a process that should take around 10 minutes.

Finally, they will proceed with the same survey for an additional 5 minutes, providing responses about their healthcare provider, patient portals, EHR errors, and some basic demographic details.

DETAILED DESCRIPTION:
This study involves an online experiment aimed at assessing patient engagement in discovering and reporting errors in Electronic Health Records (EHRs). It is being conducted by Dr. Ryan Raimi from the Information Systems Area at The University of Texas at Dallas, in collaboration with Dr. Idris Adjerid from the Business Information Technology Department at Virginia Tech, along with Dr. Anish K. Agarwal and Dr. Raina M. Merchant from the Emergency Medicine Department at the Perelman School of Medicine, University of Pennsylvania. The research involves no deception and presents no more than minimal risk to participants, similar to the risks encountered in everyday life.

Participation typically takes no more than 20 minutes and is completely confidential. To begin, participants will voluntarily consent to take part in the study. If participants agree to participate, the study process will involve the following steps:

Survey Participation: Initially, participants will complete a short survey lasting about 5 minutes, where participants will answer questions about trust, distrust, and privacy concerns.

EHR Review: Next, participants will be instructed to access their patient portal and review their EHRs, which will take approximately 10 minutes.

Final Survey: Afterward, participants will continue the same survey for another 5 minutes, answering questions about their healthcare provider, patient portals, EHR errors, and some basic demographic information.

All responses are kept confidential, and no individual participant data will be identified. The data will be aggregated and published in a summary form only. Although the study is hosted on a secure https server, there is a minimal risk of unauthorized access (e.g., by hackers). Participants' Prolific IDs will not be linked to participants' survey responses, and the investigators will not access any personally identifying information on participants' Prolific Academic profiles.

Participation is voluntary, and choosing not to participate will not affect participants' rights or benefits. Participants may withdraw from the study at any time without penalty or loss of benefits.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should have access to their patient portal
* Subjects should have checked their EHR in the past 12 months

Exclusion Criteria:

* Not having access to their patient portal
* Not having checked their EHR in the past 12 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Reviewing EHRs | From starting the initial survey through study completion, an average of 20 minutes
  Whether or not a subject reviews their EHR

SECONDARY OUTCOMES:
EHR error discovery | From starting the initial survey through study completion, an average of 20 minutes
  Whether or not the subject has discovered an error in their EHR
EHR error reporting | From starting the initial survey through study completion, an average of 20 minutes
  Whether or not the subject has reported an error in their EHR

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Raimi, PhD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- Naveen Jindal School of Management, The University of Texas at Dallas, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in this study-after de-identification-will be made available to qualified researchers upon reasonable request. This includes participant survey responses and relevant metadata (e.g., time stamps, completion status), but will exclude any personally identifying information.
  Data will be available beginning 6 months after publication of the primary results and for a period of 2 years. Requests must include a methodologically sound proposal and will be reviewed by the study investigators. Approved requests will require a data use agreement to ensure responsible use and protection of participant privacy.
  Data will be shared via a secure data repository or encrypted file transfer, depending on the nature of the request.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Start Date: 6 months after publication of the primary results End Date: 2 years after publication
Access Criteria: Qualified researchers affiliated with academic institutions, nonprofit organizations, or government agencies will be eligible to request access to the de-identified individual participant data (IPD) and supporting documentation (including the study protocol, statistical analysis plan, informed consent form, and analytic code).
  Access will be granted to researchers who submit a methodologically sound proposal outlining the intended use of the data. Proposals will be reviewed by the study's principal investigators to assess scientific merit, alignment with ethical standards, and feasibility.
  Approved researchers will be required to sign a data use agreement to ensure responsible handling of the data and protection of participant confidentiality. Upon approval, data and supporting materials will be shared via a secure online repository or encrypted file transfer.